CLINICAL TRIAL: NCT00104676
Title: A Risk-Adapted Strategy of the Use of Dose-Dense Chemotherapy in Patients With Poor-Prognosis Disseminated Non-Seminomatous Germ Cell Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Stage II or Stage III Germ Cell Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETUG 13; FRE-FNCLCC-GETUG-13/0206 (Other: UNICANCER); 2005-001072-13 (EudraCT Number)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Extragonadal Germ Cell Tumor; Teratoma; Testicular Germ Cell Tumor
Keywords: stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor; stage II extragonadal non-seminomatous germ cell tumor; stage III extragonadal non-seminomatous germ cell tumor; testicular immature teratoma; testicular mature teratoma; adult teratoma
MeSH Terms: conditions — Teratoma; Testicular Germ Cell Tumor; Testicular Neoplasms; Carcinoma, Embryonal; Endodermal Sinus Tumor | interventions — Bleomycin; Cisplatin; Etoposide; Ifosfamide; Oxaliplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Phase 3 trial with direct individual benefit, randomized, open-label, multicenter, parallel groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Active Comparator): Patients receive 4 courses of bleomycin, etoposide, and cisplatin (BEP).
  Interventions: Biological: bleomycin sulfate; Drug: cisplatin; Drug: etoposide
- Arm II (Experimental): Patients receive 1 course of bleomycin, etoposide, and cisplatin (BEP). Patients then receive dose-dense sequential combination chemotherapy comprising cisplatin, etoposide, bleomycin, paclitaxel, oxaliplatin, and ifosfamide.
  Interventions: Biological: bleomycin sulfate; Drug: cisplatin; Drug: etoposide; Drug: ifosfamide; Drug: oxaliplatin; Drug: paclitaxel

INTERVENTIONS:
Biological: bleomycin sulfate — At least one course administered
Drug: cisplatin — At least one course administered
Drug: etoposide — At least one course administered
Drug: ifosfamide — Given in a dose-dense sequential fashion
  Arms: Arm II
Drug: oxaliplatin — Given in a dose-dense sequential fashion
  Arms: Arm II
Drug: paclitaxel — Given in a dose-dense sequential fashion
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This randomized phase III trial is comparing two different combination chemotherapy regimens to see how well they work in treating patients with stage II or stage III non-seminomatous germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare progression-free survival rates of patients with poor prognosis stage II or III non-seminomatous germ cell tumors with an unfavorable decrease of tumor markers after treatment with 1 course of bleomycin, etoposide, and cisplatin followed by subsequent treatment with 3 additional courses of bleomycin, etoposide, and cisplatin OR dose-dense sequential combination chemotherapy.
* Compare overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study.

Patients receive 1 course of bleomycin, etoposide, and cisplatin (BEP). Patients with a favorable decrease of tumor markers after 1 course of BEP receive 3 additional courses of BEP. Patients with an unfavorable decrease of tumor markers after 1 course of BEP are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive 3 additional courses of BEP.
* Arm II: Patients receive dose-dense sequential combination chemotherapy comprising cisplatin, etoposide, bleomycin, paclitaxel, oxaliplatin, and ifosfamide.

PROJECTED ACCRUAL: A total of 260 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-seminomatous germ cell tumors (NSGCT) as evidenced by 1 of the following criteria:

  * Histologically confirmed NSGCT
  * Clinical evidence of disease AND high serum human chorionic gonadotropin (HCG) or alpha-fetoprotein (AFP) levels
* Clinical stage II-III disease (disseminated disease)
* Testicular, retroperitoneal, or mediastinal primary site
* Poor prognosis disease, meeting 1 of the following criteria:

  * Mediastinal primary site
  * Non-pulmonary visceral metastases
  * One of the following lab values:

    * HCG > 50,000 UI/L
    * AFP > 10,000 ng/mL
    * Lactate dehydrogenase > 10 times upper limit of normal (ULN)

PATIENT CHARACTERISTICS:

Age

* Over 16

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine clearance > 60 mL/min

Other

* No other prior malignancy except basal cell skin cancer
* No HIV positivity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2003-11-26 (Actual); Primary Completion 2012-03-29 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (24):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States
- France (22):
  - Centre Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - C.H.U. de Brest, Brest
  - Centre Regional Francois Baclesse, Caen
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Tenon, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier de Rodez, Rodez
  - Centre Henri Becquerel, Rouen
  - CRLCC Nantes - Atlantique, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- National Cancer Institute - Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Fizazi K, Le Teuff G, Flechon A, Pagliaro L, Mardiak J, Geoffrois L, Laguerre B, Chevreau C, Delva R, Rolland F, Theodore C, Roubaud G, Gravis G, Eymard JC, Cancel M, Juzyna B, Reckova M, Naoun N, Logothetis C, Culine S. Personalized Chemotherapy on the Basis of Tumor Marker Decline in Poor-Prognosis Germ-Cell Tumors: Updated Analysis of the GETUG-13 Phase III Trial. J Clin Oncol. 2024 Oct;42(28):3270-3276. doi: 10.1200/JCO.23.01960. Epub 2024 Aug 21. PMID 39167741
- [Derived] Fizazi K, Pagliaro L, Laplanche A, Flechon A, Mardiak J, Geoffrois L, Kerbrat P, Chevreau C, Delva R, Rolland F, Theodore C, Roubaud G, Gravis G, Eymard JC, Malhaire JP, Linassier C, Habibian M, Martin AL, Journeau F, Reckova M, Logothetis C, Culine S. Personalised chemotherapy based on tumour marker decline in poor prognosis germ-cell tumours (GETUG 13): a phase 3, multicentre, randomised trial. Lancet Oncol. 2014 Dec;15(13):1442-1450. doi: 10.1016/S1470-2045(14)70490-5. Epub 2014 Nov 13. PMID 25456363

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 263 patients registered 255 were evaluated for biomarker decrease after one cycle of BEP. Eight patients were not evaluated for biomarker decrease: 6 patients died early, 1 patient 1 withdrew consent and 1 patient was included by error. 1 patient was not covered by EC approval and excluded froma analysis. The 203 patients with unfavorable decrease in tumor biomarkers were randomized in Arm I (98 patients) or Arm II (105 patients).
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 98 | 105
Completed | 91 | 91
Not Completed | 7 | 14
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — treatment interruption | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 98 | 105 | 203
Age, Continuous [Median (Full Range); unit: Years] | 27 [17 to 65] | 30 [16 to 51] | 30 [16 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 98 | 105 | 203
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
  Slovakia | 9 | 9 | 18
  France | 79 | 87 | 166

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate After 1 Course of Treatment
Description: Primary objective is to compare the progression-free survival of participants after 1 cycle of treatment, treated randomly by 3 additional cycles of BEP (Arm I) or by T-BEP-Oxaliplatin/cisplatin-ifosfamide-Bleomycin (Arm II). The median progression-free survival rate was defined as the median percentage of participants alive without disease progression after 1 course of treatment.
Time Frame: 3 years from randomization
Population: The primary endpoint for the study was the comparison of the PFS rates in the population of participants with a poor prognostic non-seminomatous germ cell tumors and with an unfavorable decrease in tumor biomarkers, randomized to either Unfav-BEP Control Arm (Arm I) or Unfav-Dose-Dense Arm (Arm II).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 98 | 105
percentage of participants | 48 [38 to 59] | 59 [49 to 68]
Statistical Analysis 1: Comparison: Arm I vs Arm II; To detect an absolute difference of 20% in progression-free survival at 3-years between Arm I and Unfav-Dose-Dense Arm II (46% versus 66%) with the possibility that 80 events (progressive disease and death) may be observed during this period, a total of 196 participants, 98 per group needed to be included, with an additional 25% of patients for a total of 260 participants required; Test type: Superiority; p = 0.05, Log Rank; Adjusted on the stratification factor (treatment centers); Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.44 to 1.00]

2. Secondary Outcome: Overall Survival
Description: To evaluated the overall survival in both groups in participants presenting fast and slow decrease in serum levels of tumor markers. The median overall survival was defined as the median percentage of participants alive after 1 course of treatment.
Time Frame: 3 years from randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 98 | 105
percentage of participants | 65 [55 to 75] | 73 [64 to 81]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority; p = 0.34, Log Rank; Adjusted on the stratification factor (treatment centers); Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.46 to 1.31]

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II
All-Cause Mortality (participants affected / at risk) | 61/98 | 66/105
Serious Adverse Events (participants affected / at risk) | 37/98 | 58/105
Other Adverse Events (participants affected / at risk) | 98/98 | 105/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=98) | Arm II (N=105)
Acute leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 7
Aplasia bone marrow (Blood and lymphatic system disorders) | 3 | 2
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Febrile aplasia (Blood and lymphatic system disorders) | 1 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 9
Myeloid leukemia, acute (Blood and lymphatic system disorders) | 4 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Myelodysplasia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 26 | 17
Neutropenia aggravated (Blood and lymphatic system disorders) | 2 | 2
Neutropenia malignany (Blood and lymphatic system disorders) | 0 | 1
Thrombopenia (Blood and lymphatic system disorders) | 1 | 7
Pericarditis (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Fistula of small intestine (Gastrointestinal disorders) | 1 | 0
Anal abscess (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Mucositis (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Fever (General disorders) | 3 | 5
Catheter infection (Injury, poisoning and procedural complications) | 4 | 3
Catheter blocage (Injury, poisoning and procedural complications) | 0 | 1
General physical health deterioration (Gastrointestinal disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 2
Liver damage (Hepatobiliary disorders) | 0 | 3
Infection (Infections and infestations) | 1 | 6
scrotal abscess (Infections and infestations) | 1 | 0
Septicemia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 5
vomiting post chemotherapy (Injury, poisoning and procedural complications) | 0 | 1
weight decrease (Investigations) | 0 | 1
Liver enzyme abnormal (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes with renal manifestations (Metabolism and nutrition disorders) | 0 | 1
Gout acute (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 1
Inguinal abscess (Musculoskeletal and connective tissue disorders) | 0 | 1
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Mediastinal neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Coma (Nervous system disorders) | 1 | 0
Convulsions (Nervous system disorders) | 1 | 0
Hypertension intracranial (Nervous system disorders) | 1 | 0
Consciousness loss of (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 5
Paraesthesia (Nervous system disorders) | 0 | 3
Polyneuropathy toxic (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 6
Stroke (Nervous system disorders) | 0 | 1
Anxiety depression (Psychiatric disorders) | 0 | 1
Ureteral stricture (Renal and urinary disorders) | 1 | 1
Renal insufficiency (Renal and urinary disorders) | 0 | 4
Renal failure acute (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstruction lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Platelet transfusion (Surgical and medical procedures) | 1 | 0
Cutaneous hypersensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal aortic aneurysm (Vascular disorders) | 1 | 0
Epistaxis (Vascular disorders) | 1 | 0
Intracerebral hemorrhage (Vascular disorders) | 0 | 1
Peritoneal haemorrhage (Vascular disorders) | 0 | 1
Phlebitis lower limb (Vascular disorders) | 0 | 1
Tumor hemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=98) | Arm II (N=105)
Rash (Skin and subcutaneous tissue disorders) | 18 | 27
Nausea (Gastrointestinal disorders) | 72 | 91
Diarrhea (Gastrointestinal disorders) | 20 | 52
Mucositis (Gastrointestinal disorders) | 18 | 45
Liver function test increased (Hepatobiliary disorders) | 43 | 36
Neuropathy (Nervous system disorders) | 21 | 82
Auditory disorder (Ear and labyrinth disorders) | 28 | 52
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 | 43
Creatinine (Hepatobiliary disorders) | 9 | 29
Asthenia (General disorders) | 76 | 90
Infection (Infections and infestations) | 23 | 33
Hemoglobin (Blood and lymphatic system disorders) | 98 | 105
Granulocytes (Blood and lymphatic system disorders) | 79 | 84
Platelets (Blood and lymphatic system disorders) | 72 | 88
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No